CLINICAL TRIAL: NCT00006225
Title: Ex Vivo Expanded Megakaryocytes for Supportive Care of Breast Cancer Patients: A Phase I/II Study
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Breast Cancer or Hematologic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NU 97B2; NU-97B2; NCI-V00-1611
Record Dates: First submitted 2000-09-11; First posted 2003-05-07 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic/Myeloproliferative Diseases
Keywords: stage IV adult Hodgkin lymphoma; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent adult Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system lymphoma; male breast cancer; intraocular lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; chronic myelomonocytic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Breast Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic-Myeloproliferative Diseases; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Breast Neoplasms, Male; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; flt3 ligand protein; Thrombopoietin; Stem Cell Factor

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant flt3 ligand
Biological: recombinant human thrombopoietin
Biological: recombinant interleukin-3
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy.

PURPOSE: Randomized phase I/II trial to study the effectiveness of peripheral stem cell transplantation in treating patients who have breast cancer or hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of ex vivo expanded megakaryocytes (EVE MK) as a supplement to peripheral blood stem cell (PBSC) transplantation in patients with breast cancer or hematologic malignancies.
* Compare the effect of this treatment regimen on platelet recovery and platelet function in these patients vs historical controls.
* Compare the frequency of malignant cells in the EVE MK vs the uncultured PBSC collection in these patients.
* Determine the optimal time of MK harvest for the production of platelets in vivo.
* Determine the required number of MKs for clinical efficacy in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 durations of CD34+ culture times (6 days vs 9 days).

After an initial harvest of filgrastim (G-CSF)-mobilized autologous peripheral blood stem cells (PBSC) for transplantation, patients receive one additional dose of G-CSF and undergo one additional apheresis. The CD34+ cells are cultured in the presence of recombinant human thrombopoietin, interleukin-3, and flt3 ligand to expand megakaryocytes. Patients then undergo treatment with high-dose chemotherapy (and, in some cases, total body irradiation) followed by reinfusion of the conventional PBSC harvest and the ex vivo expanded megakaryocytes.

Patients are followed until blood counts recover.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of carcinoma of the breast or hematologic malignancies
* No metastases to bone marrow
* Planned high-dose chemotherapy with autologous peripheral blood stem cell transplantation
* At least 2.0 million CD34+ cells/kg collected
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 60

Sex:

* Female or male

Menopausal status:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* SGOT or SGPT less than 2.5 times upper limit of normal (ULN)
* Bilirubin less than 2.5 times ULN (except in Gilbert's syndrome)
* Alkaline phosphatase less than 2.5 times ULN
* No active hepatitis B or C

Renal:

* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* Normal ejection fraction

Pulmonary:

* DLCO at least 50% predicted
* FEV_1 and/or FVC at least 75% predicted

Other:

* No concurrent serious nonneoplastic disease that would preclude study entry
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-11; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States